CLINICAL TRIAL: NCT00265993
Title: The Efficacy of Subcutaneous Enoxaparin Once Daily in the Treatment of Acute Venous Thromboembolic Disease: an Open-labelled, Non-comparative, Multicentric, Phase IV Trial
Brief Title: Enoxaparin in Acute Venous Thromboembolic Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP4563A_4001
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Enoxaparin

ARMS (1):
- 1 (Experimental): enoxaparin
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: enoxaparin — * All patients will be treated with enoxaparin 1.5 mg/kg, once a day, subcutaneously for up to 10 days.
  * Long-term oral anticoagulation will be started in all patients after 24 hours of initiation of enoxaparin treatment and continued at least for 3 months.

SUMMARY:
Study objectives :

* To evaluate the efficacy/safety profile of enoxaparin once a day treatment in acute venous thromboembolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic lower-extremity deep venous thrombosis confirmed by doppler USG (ultrasonography), with or without confirmed symptomatic pulmonary embolism associated with provoked risk factors

Exclusion Criteria:

* Patients with a history of heparin or warfarin treatment longer than 24 hours,
* Patients requiring thrombolytic treatment,
* Patients having thrombophilia diagnosis,
* Patients with prior deep vein thrombosis or pulmonary emboli evidence,
* Patients with familial bleeding disorder,
* Patients who are at any known bleeding risk, such as active bleeding, active ulcerative bowel disease, angiodysplasia and having oculary, spinal or central nervous system surgery within the last month
* Patients with renal failure (serum creatinine concentration > 180 mmol/L or > 2.03 mg/dL),
* Patients with severe hepatic failure
* Patients with history of allergy against heparin and protamine,
* Patients with history of thrombocytopenia associated with heparin administration or of skin necrosis after heparin or warfarin treatment,
* Patients participating in another clinical study within the last 4 months
* Patients who are pregnant

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2004-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Frequency of bleeding emerged during the study drug administration; Frequency of bleeding emerged during 3 months of monitorization when the patient is on oral anticoagulants. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)